CLINICAL TRIAL: NCT07160088
Title: Delayed Ischemic Neurological Deficit in Patients With Aneurysmal Subarachnoid Hemorrhage: Real World Study (DINDaSAH)
Brief Title: DIND in Patients With aSAH : Real World Study
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Lidan Jiang, Principal Investigator, Xuanwu Hospital, Beijing
Other Study IDs: [2025]264-002
Record Dates: First submitted 2025-08-14; First posted 2025-09-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage (aSAH)
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — This is an observational study without study-related intervention. All the treatments will be depended on the attending doctors and according to the related guidelines.

SUMMARY:
In recent years, with the active application of clinical monitoring and treatment methods, the survival rate of patients with aneurysmal subarachnoid hemorrhage (SAH) has improved, but still a certain proportion of patients develop chronic and disabling neurological deficits, namely delayed ischemic neurological deficits (DIND). The incidence of DIND is not clear, and the causes are diverse. Symptomatic vasospasm is only one of the possible causes, and early diagnosis is difficult. Up to now, there is no gold standard for diagnosis and no relevant treatment guidelines.

Given these reasons, this study intends to conduct a prospective multicenter observational study to collect relevant information on diagnostic methods (neurological symptoms in clinical examinations or changes in monitoring by instruments) and treatment methods, describe the incidence of delayed cerebral ischemia (DIND) in patients with subarachnoid hemorrhage (SAH), evaluate the different treatment strategies adopted by participating centers, and compare these strategies in terms of mortality and short-term and long-term neurological outcomes, and describe the indications, usefulness, and treatment intensity of intracranial pressure monitoring of the brain parenchyma during SAH in patients.

Study design: This study is a multicenter, prospective, observational study. The study subjects are patients with subarachnoid hemorrhage as the primary diagnosis, admitted to the intensive care unit and receiving treatment. The treatment of patients with subarachnoid hemorrhage (SAH) and delayed cerebral ischemia (DIND) is the responsibility of the professional medical and surgical teams of each center.

Study period: The enrollment period is 12 months from the start of ethical approval, and the follow-up period is 12 months after the onset.

Inclusion criteria:

① Age ≥ 18 years; ② Aneurysmal subarachnoid hemorrhage (confirmed by DSA/CTA); ③ Admitted to the intensive care unit; ④ Signed informed consent.

Exclusion criteria:

① Unidentified cause of subarachnoid hemorrhage (no visible aneurysm); ② Traumatic SAH; ③ Complicated with brain tumors or arteriovenous malformations.

Endpoints:

Primary endpoints: The occurrence of suspected DIND: Whether it is indicated by neurological clinical examination (such as the patient being conscious or in a light sedated state), or by the monitoring of instruments (if clinical examination is impossible), suggesting the possibility of DIND, regardless of whether there is imaging confirmation or not, can be considered as suspected DIND.

Secondly endpoints: - The clinical application of diagnostic and monitoring methods in the identification and management of DIND in patients with aSAH.

* Evaluation of mortality and neurological functional prognosis (GOSE and mRS) at 6 months and 12 months after onset.
* Comparison of changes in intracranial pressure (ICP) in patients with ICP monitoring and the intensity of the treatment received (Therapy Intensity Level, TIL).

Sample size:

The enrollment will be as much as possible during the enrollment period (totally approximately 1000 cases).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Primary diagnosis of subarachnoid hemorrhage due to rupture of a cerebral artery aneurysm confirmed by cerebral angiotomography or intracranial vessel angiography, requiring admission to the Intensive Care Unit (ICU).
3. Signature of the Informed Consent Form for participation in the study in accordance with local applicable regulations.

Exclusion Criteria:

1. Age < 18 years old
2. Primary diagnosis of subarachnoid hemorrhage withouth a visible aneurysm, i.e., post-traumatic or caused by an arteriovenous malformation or bleeding from a brain tumor.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will enroll all the adult aSAH patients admitted in the Intensive Care Units (ICU) of several hospitals located in China, who meet the inclusion/exclusion criteria of this study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DIND in patients with SAH, where-after excluding other possible causes such as hydrocephalus, seizures, rebleeding, and hyponatremia. | From Day 1 to one month
  In a patient who is awake or can be awakened to undergo a clinical neurological examination, DIND is diagnosed when there is evidence of either: a focal neurological deterioration (at least one of the following: hemiparesis, aphasia, hemianopsia, or neglect), or a global deterioration (sudden neurological worsening resulting in a decrease of at least two points on the GCS or on the NIHSS, or the appearance of anisocoria or non-reactive pupils).
  In comatose or non-awakable patients, DIND is diagnosed when at least one of the following alterations is observed:
  NPi: <3 on a scale from 0 to 5 TCD:vasospasm of a major cerebral artery CEEG:presence of reduced alpha variability and/or a decreased α/δ ratio, or the appearance of depolarization waves in clusters of 2-5 mm/min PbtO2:<20 mmHg CTP:ischemic core or penumbra, or <15 ml/100g/min DSA:reduction of ≥50% in the diameter of a major cerebral artery CT/MRI:presence of ischemic lesion

SECONDARY OUTCOMES:
Mortality and neurological-functional outcomes (GOSE - Glasgow Outcome Scale Extended) at 6 and 12 months after the acute event | from Day 1 to follow-up at 12 months
  In Glasgow Outcome Scale Extended (GOSE), the minimum is 1(dead) and maximum 8 (Good recovery, near complete), higher scores mean a better outcome.
Mortality and neurological-functional outcomes (mRS - modified Rankin Scale) at 6 and 12 months after the acute event | from Day 1 to follow-up at 12 months
  In mRS (modified Rankin Scale), the minimum is 0 (complete recovered), and maximum 6 (dead), higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Capital Medical University, Beijing, Beijing Municipality, China